CLINICAL TRIAL: NCT03281889
Title: Craniospinal Irradiation Using Proton Beam Scanning With Selective Vertebral Body/Bone Sparing to Improve Marrow Reserve and Decrease Growth Decrement for Children
Brief Title: Proton Craniospinal Irradiation With Bone Sparing to Decrease Growth Decrement From Radiation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kevin X. Liu, MD, DPHIL, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-283; U19CA021239-37 (NIH)
Record Dates: First submitted 2017-09-08; First posted 2017-09-13 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Brain Tumor
Keywords: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms | interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Proton Radiotherapy (Experimental): * Patients will be treated with Proton Beam once daily 5 days per week.
  * Doses will be prescribed such that maximum possible coverage is achieved
  Interventions: Radiation: Proton Beam

INTERVENTIONS:
Radiation: Proton Beam — precision radiation that reduce the negative effects radiation has on the surrounding non-cancerous growing and developing tissue

SUMMARY:
This research study is studying proton radiation as a possible treatment for brain tumor that requires radiation.

The radiation involved in this study is:

-Proton Radiation

DETAILED DESCRIPTION:
This research study is a Pilot Study to determine whether using proton therapy in participants that require craniospinal radiation (whole brain and spinal cord radiation therapy) with sparing of the bony spine will work. This is the first time investigators are examining bone sparing proton therapy in pediatric craniospinal radiation.

The FDA (the U.S. Food and Drug Administration) has not approved proton radiation for this specific disease but it has been approved for other uses.

In this research study, the investigators are studying proton radiation in participants that require craniospinal radiation. The standard of care for this procedure is photon radiation, which is very similar to proton radiation. The investigators believe that the precision of proton radiation may help to reduce the negative effects radiation has on the surrounding non-cancerous growing and developing tissue

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 3 years and ≤ 18 years at the time of registration
* Histologically proven malignancy necessitating cranio-spinal irradiation. This will include patients with a diagnosis of medulloblastoma, Supratentorial primitive neuroectodermal tumor (SPNET), germ cell tumor (GCT), disseminated ependymoma, embryonal tumor with abundant neuropil and true rosettes (ETANTR), Atypical Teratoid/Rhabdoid Tumor (ATRT), and disseminated low-grade glioma (LGG).
* Life expectancy ≥ 12 months.
* Signed informed consent document and assent when appropriate.
* HGB of > 10 g/L and PLT count > 80 K/uL

Exclusion Criteria:

* Any prior therapeutic radiation therapy > 500 cGy has been delivered.
* Individuals with a history of a different malignancy are ineligible except for the following circumstances: if they have been disease-free for at least 5 years and are deemed by the investigator to be a low-risk for recurrence of that malignancy; or, have had only cervical cancer in situ, or basal cell or squamous cell carcinoma of the skin.
* Any major uncontrolled or poorly controlled intercurrent illness that would limit compliance with study requirements.
* Pregnant females are excluded. Females of childbearing age/menstruating must confirm that either they are not sexually active or have a negative pregnancy test prior to initiation of radiation therapy.
* Patients that receive concurrent chemotherapy with the exception of concurrent Vincristine.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of cranio-spinal irradiation (CSI) utilizing intensity-modulated proton therapy (IMPT) with pencil beam scanning (PBS) for vertebral body sparing (VBS) in pediatric patients. | 3 months
  IMPT using PBS delivery will be considered to be feasible as a VBS technique for CSI in pediatric patients if the rate of grade 3/4 hematologic toxicity were no more than 5% within 3 months after the completion of radiation treatment, within the range associated with conventional techniques of CSI. Toxicity will be assess using Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.

SECONDARY OUTCOMES:
Early marrow changes in the vertebral bodies | 2 years
  Summary of early marrow changes in the vertebral bodies by Magnetic resonance imaging (MRI) of the spine during radiation therapy (RT) by comparing one study MRI to the baseline pre-RT MRI.
Vertebral column growth (measured by MRI) over 1 year | Last day of treatment to 1 year later
  Summary of vertebral column growth (measured by MRI) over 1 year following vertebral body sparing cranio-spinal irradiation in pediatric patients.
Change in sitting height and standing height | Annually for 5 years
  Summary of the changes in the participants sitting and standing heights.
Time to abnormality in spinal curvature | 5 years
  Participants are monitored both clinically and by MRI for any abnormality in spinal curvature. The time to abnormality in spine curvature will be measured from the start of radiation to the date of documented abnormality or censored at the date of last follow-up for patients still alive with normal spine.
Disease Free Survival | 5 years
  Disease-free survival is measured from the start of radiation to the date of progressive disease based on imaging studies obtained as standard care or to the date of death due to any cause, whichever is earlier. Disease-free survival will be estimated using the Kaplan-Meier method. Patients without progressive disease and still alive will be censored at their date of last contact.
Pattern of Disease Relapse | 2 years
  Summary of the sites where the cancer relapses. Relapse is the regrowth of cancer cells.
Complete blood counts (CBC) over time | Annually for 5 years
  Summary of the change in complete blood counts (CBC) over time as determined by yearly blood samples.
Change in levels of vitamin D, calcium, and growth hormones over time | Annually for 5 years
  Summary of the changes in blood levels of vitamin D, calcium, and growth hormones.
Weight | Annually for 5 years
  Summary of the changes in weight of the participants as assessed by yearly evaluations.
BMI | Annually for 5 years
  Summary of the body mass index (BMI) of the participants as assessed by yearly physical evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon MacDonald, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No